CLINICAL TRIAL: NCT01691742
Title: Double-Blind Randomized Controlled Trial of MiraLAX Versus Placebo to Prevent Constipation Following Urogynecologic Surgery in Women Receiving Routine Docusate Sodium
Brief Title: MiraLAX Versus Placebo to Prevent Constipation Following Urogynecologic Surgery
Acronym: MVP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: American Urogynecologic Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro00035126
Record Dates: First submitted 2012-09-18; First posted 2012-09-25 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2014-10

CONDITIONS: Post Procedural Constipation
Keywords: Postoperative constipation; Urogynecologic Surgery; MiraLax; Docusate Sodium
MeSH Terms: interventions — polyethylene glycol 3350; maltodextrin; Magnesium Hydroxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo maltodextrin 17g powder daily for 5 days postoperatively following urogynecologic surgery
  Interventions: Drug: Placebo; Drug: Rescue Laxative
- MiraLax (Active Comparator): MiraLax 17g powder daily for 5 days postoperatively following urogynecologic surgery
  Interventions: Drug: MiraLax; Drug: Rescue Laxative

INTERVENTIONS:
Drug: MiraLax — MiraLax 17g powder daily for 5 days postoperatively following urogynecologic surgery
  Other Names: PEG 3350; Polyethylene Glycol 3350
  Arms: MiraLax
Drug: Placebo — Placebo maltodextrin 17g powder daily for 5 days postoperatively following urogynecologic surgery
  Other Names: Maltodextrin
  Arms: Placebo
Drug: Rescue Laxative — All participants will be instructed to take Milk of Magnesia with standard over-the-counter dosing as a recue laxative if the subject has not had a bowel movement by postoperative day 6.
  Other Names: Milk of Magnesia

SUMMARY:
A. Purpose To compare MiraLAX versus placebo for preventing constipation in the immediate postoperative period following pelvic reconstructive surgery in women taking routine docusate sodium.

B. Objectives

1. Specific Aims Specific Aim 1: To compare time to first bowel movement (BM) between MiraLAX versus placebo in women receiving routine docusate sodium after pelvic reconstructive surgery.

   Specific Aim 2: To compare patient reported outcomes of BM quality and associated gastrointestinal (GI) symptoms between MiraLAX versus placebo using the Bristol stool scale and the validated Patient Assessment of Constipation Symptom Questionnaire (PAC-SYM) in women receiving routine docusate sodium after pelvic reconstructive surgery.

   Specific Aim 3: To evaluate GI-related quality of life between MiraLAX versus placebo utilizing the validated Patient Assessment of Constipation Quality-of-Life Questionnaire (PAC-QOL) in women receiving routine docusate sodium after pelvic reconstructive surgery.
2. Hypotheses The investigators hypothesize that MiraLAX will optimally prevent constipation following pelvic reconstructive surgery by decreasing time to first BM, decreasing GI symptoms associated with constipation, and increasing measures of GI-related quality of life, while minimizing the bothersome side effects associated with stimulant laxatives.

DETAILED DESCRIPTION:
This is a randomized double-blind placebo-controlled clinical trial of MiraLAX versus placebo in women undergoing pelvic reconstructive surgery receiving routine docusate sodium. Subjects will be screened for eligibility during their preoperative visits and once enrolled, they will be randomized to receive MiraLAX or placebo starting on postoperative day (POD) 1 and continuing through POD 5. Subjects will be instructed to stop taking this medication if they experience any diarrhea. Subjects in both arms will be instructed to take milk of magnesia as a rescue laxative if they do not experience a BM by the morning of POD 6. All subjects will be provided a 30 day supply of docusate sodium and be instructed to begin this medication on POD 1.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking female patients
* > 18 years of age
* Not pregnant (patients of childbearing potential will have a serum pregnancy test done pre-operatively as part of their surgical planning)
* Undergoing surgery for pelvic organ prolapse or stress urinary incontinence
* Recruited from the Duke University Division of Urogynecology

Exclusion Criteria:

* Allergy/hypersensitivity to study medications
* Cardiac or renal disease
* Takes chronic daily laxatives
* Excluded if unable to complete at least 5 days of a 7 day baseline bowel diary
* Excluded if mesh resection or Interstim procedure
* Excluded if concurrent surgery includes anal sphincteroplasty or rectovaginal fistula repair

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2012-09; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Time to first postoperative bowel movement | First postoperative week
  The primary outcome is time to first postoperative bowel movement (in hours, converted to days) based upon postoperative bowel diary. Time will be calculated based upon date and time of first postoperative bowel movement from start time of surgery.

SECONDARY OUTCOMES:
Other postoperative medication use | First postoperative week
  Rescue laxative use, daily pain level and narcotic use will be obtained from postoperative bowel diaries.
Evaluation of symptoms and quality of life related to constipation | First postoperative week
  The investigators will evaluate BM quality based upon Bristol stool scale. Straining, abdominal or rectal pain, incomplete evacuation and the impact of these symptoms on GI-related quality of life will be assessed by the PAC-SYM and PAC-QOL validated questionnaires. The PAC-SYM is a validated 12-item questionnaire based upon the Rome criteria for constipation and is tailored to assess a change in symptoms following an intervention.2 This questionnaire has been previously used with success in studies with urogynecologic patients. The PAC-QOL is a validated 28-item questionnaire assessing quality-of-life issues, including burden of constipation on daily functioning and well-being. The Bristol stool scale, which is a visual BM rating scale from 1 to 7, provides a validated measure of gut transit time based upon the shape, consistency and appearance of BM.
Symptoms of Over-Effectiveness | First Postoperative Week
  Symptoms of over-effectiveness, including abdominal pain or cramping, bloating, loose stools, watery diarrhea and their impact on GI-related quality of life will be evaluated based upon bowel diaries, Bristol stool scales and the PAC-SYM and PAC-QOL questionnaires.
Evaluation of symptoms and quality of life related to constipation 6-weeks postoperatively | 5-7 weeks postoperatively
  The investigators will evaluate BM quality based upon Bristol stool scale. Straining, abdominal or rectal pain, incomplete evacuation and the impact of these symptoms on GI-related quality of life will be assessed by the PAC-SYM and PAC-QOL validated questionnaires. The PAC-SYM is a validated 12-item questionnaire based upon the Rome criteria for constipation and is tailored to assess a change in symptoms following an intervention.2 This questionnaire has been previously used with success in studies with urogynecologic patients. The PAC-QOL is a validated 28-item questionnaire assessing quality-of-life issues, including burden of constipation on daily functioning and well-being. The Bristol stool scale, which is a visual BM rating scale from 1 to 7, provides a validated measure of gut transit time based upon the shape, consistency and appearance of BM.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony G Visco, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Department of Urogynecology, Durham, North Carolina, United States

REFERENCES:
- [Derived] Edenfield AL, Siddiqui NY, Wu JM, Dieter AA, Garrett MA, Visco AG. Polyethylene Glycol 3350 and Docusate Sodium Compared With Docusate Sodium Alone After Urogynecologic Surgery: A Randomized Controlled Trial. Obstet Gynecol. 2016 Sep;128(3):543-9. doi: 10.1097/AOG.0000000000001565. PMID 27500338